CLINICAL TRIAL: NCT03866850
Title: Degenerative Consequences of Congenital Deafness
Status: Terminated | Type: Observational
Why Stopped: PI passed away. Ending grant and closing lab.
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Heather Wright, Professor, East Carolina University
Other Study IDs: Zhou_R01_study2
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Congenital Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cochlear implant users with late-onset deafness: Examine charge integration (Detection threshold as a function of phase duration).
  Examine neural spatial excitation patterns with long and short phase duration. Measure speech recognition using long and short phase duration stimulation patterns.
  Interventions: Behavioral: Phase duration
- Cochlear implant users with early-onset deafness: Examine charge integration (Detection threshold as a function of phase duration) and compare that with the late-onset group.
  Examine neural spatial excitation patterns with long and short phase duration within the non-leaky phase duration range.
  Measure speech recognition using long and short phase duration stimulation patterns.
  Interventions: Behavioral: Phase duration

INTERVENTIONS:
Behavioral: Phase duration — We will vary the phase duration in the stimulation, and examine detection threshold, spatial spread of neural excitation, and speech recognition as the outcomes.

SUMMARY:
In this study, the investigators will study one of the basic biophysical properties of the auditory nerve, charge integration, behaviorally (detection threshold versus phase duration functions). The investigators will compare charge integration in two subject groups: congenitally deafened and deafened at a later age in life. The investigators will then examine if behaviorally estimated neural excitation patterns differ between short phase duration and long phase duration stimulation. Lastly, The investigators will measure if speech recognition improves with using long phase duration stimulation, relative to using the standard default short phase duration stimulation. The primary endpoint of the study is speech recognition, and the secondary endpoints are the steepness of the detection threshold versus phase duration functions, and the width of psychophysically estimated neural excitation.

ELIGIBILITY:
Inclusion Criteria:

* Cochlear Nucleus cochlear implant users or Advanced Bionics cochlear implant users
* Native speakers of English
* Early onset of deafness (< 3 years of age); no requirement for age at implantation
* Late onset of deafness (> 3 years of age); matched in duration of deafness to the early onset group
* Has had device experience for at least one year
* Can be child or adult at the time of enrollment

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with cochlear implants (Advanced Bionics and Cochlear Nucleus devices)
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Slope of the strength duration function | starting 6 months post award notice and will take up to 4 years to complete
  Subjects will be measured for detection thresholds as a function of phase duration of the pulse train and the slope of the function will be derived.

SECONDARY OUTCOMES:
Psychophysically estimated neural excitation width | starting 6 months post award notice and will take up to 4 years to complete
  Subjects will be measured for psychophysical forward-masked spatial tuning curves using stimuli with long and short phase duration.
Speech recognition using long phase duration | starting 6 months post award notice and will take up to 4 years to complete
  Subjects' speech recognition performance will be evaluated using CUNY and TIMIT sentences with long and short phase duration stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Communication Sciences and Disorders, ECU, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hancock KE, Chung Y, Delgutte B. Congenital and prolonged adult-onset deafness cause distinct degradations in neural ITD coding with bilateral cochlear implants. J Assoc Res Otolaryngol. 2013 Jun;14(3):393-411. doi: 10.1007/s10162-013-0380-5. Epub 2013 Mar 5. PMID 23462803
- [Background] Hancock KE, Noel V, Ryugo DK, Delgutte B. Neural coding of interaural time differences with bilateral cochlear implants: effects of congenital deafness. J Neurosci. 2010 Oct 20;30(42):14068-79. doi: 10.1523/JNEUROSCI.3213-10.2010. PMID 20962228
- [Background] Hardie NA, Shepherd RK. Sensorineural hearing loss during development: morphological and physiological response of the cochlea and auditory brainstem. Hear Res. 1999 Feb;128(1-2):147-65. doi: 10.1016/s0378-5955(98)00209-3. PMID 10082295
- [Background] Leake PA, Snyder RL, Rebscher SJ, Moore CM, Vollmer M. Plasticity in central representations in the inferior colliculus induced by chronic single- vs. two-channel electrical stimulation by a cochlear implant after neonatal deafness. Hear Res. 2000 Sep;147(1-2):221-41. doi: 10.1016/s0378-5955(00)00133-7. PMID 10962187
- [Background] McKay CM. Forward masking as a method of measuring place specificity of neural excitation in cochlear implants: a review of methods and interpretation. J Acoust Soc Am. 2012 Mar;131(3):2209-24. doi: 10.1121/1.3683248. PMID 22423717
- [Background] Rattay F. Analysis of models for extracellular fiber stimulation. IEEE Trans Biomed Eng. 1989 Jul;36(7):676-82. doi: 10.1109/10.32099. PMID 2744791
- [Background] Sharma A, Gilley PM, Dorman MF, Baldwin R. Deprivation-induced cortical reorganization in children with cochlear implants. Int J Audiol. 2007 Sep;46(9):494-9. doi: 10.1080/14992020701524836. PMID 17828665
- [Background] Svirsky MA, Robbins AM, Kirk KI, Pisoni DB, Miyamoto RT. Language development in profoundly deaf children with cochlear implants. Psychol Sci. 2000 Mar;11(2):153-8. doi: 10.1111/1467-9280.00231. PMID 11273423
- [Background] Teoh SW, Pisoni DB, Miyamoto RT. Cochlear implantation in adults with prelingual deafness. Part II. Underlying constraints that affect audiological outcomes. Laryngoscope. 2004 Oct;114(10):1714-9. doi: 10.1097/00005537-200410000-00007. PMID 15454759
- [Background] Trune DR. Influence of neonatal cochlear removal on the development of mouse cochlear nucleus: I. Number, size, and density of its neurons. J Comp Neurol. 1982 Aug 20;209(4):409-24. doi: 10.1002/cne.902090410. PMID 7130465
- [Background] van den Honert C, Stypulkowski PH. Physiological properties of the electrically stimulated auditory nerve. II. Single fiber recordings. Hear Res. 1984 Jun;14(3):225-43. doi: 10.1016/0378-5955(84)90052-2. PMID 6480511
- [Background] Kong YY, Deeks JM, Axon PR, Carlyon RP. Limits of temporal pitch in cochlear implants. J Acoust Soc Am. 2009 Mar;125(3):1649-57. doi: 10.1121/1.3068457. PMID 19275322